CLINICAL TRIAL: NCT04113395
Title: Concordance and Accuracy of Magnetic Resonance Imaging in the Detection of Meningiomas: Optimizing Sequences With Low Doses of Gadolinium
Brief Title: Concordance and Accuracy of MRI in the Detection of Meningiomas: Optimizing Sequences With Low Doses of Gadolinium
Acronym: CAMOMILLE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2019_14
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sequences T1 FE — T1 TSE and T1 TFE sequences with a duration of 6 minutes are added to the imaging protocol.
  Other Names: T1 TFE sequences

SUMMARY:
Meningioma, an extra-axial brain tumor developed at the expense of meninges, accounts for 35% of central nervous system tumors, and its incidence is estimated at 3% in large autopsy series.

The current gold standard for screening and monitoring cerebral meningiomas is MRI with injection of gadoline-contrast product. However, the use of some of these products is problematic, due to gadolinium deposits observed in patients who have had several injections during their lifetime, especially in patients followed for multiple sclerosis.

Recently, the French National Agency for the Safety of Medicines and Health Products (ANSM) issued recommendations concerning the screening of meningiomas in patients at risk, particularly in people treated with cyproterone acetate. It is a synthetic progestogen steroid with anti-androgenic properties. It is used to treat hyperandrogenic syndromes in women or in the palliative treatment of prostate cancer in men. Its long-term use seems to be associated with a significant over-risk of developing meningiomas, brain tumours affecting meninges. This increased risk is multiplied by 7 in women exposed to high doses of cyproterone acetate, and by 20 over a cumulative dose of 60 grams, or about 5 years of treatment at 50 mg/day or 10 years at 25 mg/day. The ANSM recommends that a cerebral MRI be performed at the beginning of treatment for all patients, as well as a control MRI renewed at 5 years and then every 2 years if the MRI at 5 years is normal. These recommendations will lead to a large number of MRIs involving an injection of contrast agent in this population, with potential immediate or delayed serious adverse effects.

New techniques, such as Arterial Spin Labelling (ASL), or black blood sequences optimized for contrast detection, have been developed. These could detect meningeal anomalies and more particularly meningiomas without contrast injection, or with a significantly lower dose of contrast agent.

These techniques have not been specifically studied for screening or monitoring meningeal lesions, but it seems relevant and important to be able to validate protocols that reduce gadolinium doses given the high number of screening and follow-up MRIs in the general population.

Patients presenting for brain MRI screening or meningioma follow-up will have the usual MRI sequences for their management, and the sequences performed at 1/6th of the standard dose of Gadolinium that are added for research. These new sequences will add approximately 6 minutes of additional examination time.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient performing MRI as part of a screening or follow-up of known meningioma
* Express consent to participate in the study

Exclusion Criteria:

* Contraindication for MRI (electrical device, metallic foreign body, claustrophobia)
* Known hypersensitivity to the contrast medium (Gadolinium)
* Known renal failure: glomerular filtration rate <30mL/min
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the radiology department of the Adolphe de Rothschild Foundation for an MRI, as part of a screening or monitoring of meningioma
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic concordance in terms of meningioma detection between the 3T MRI sequences with a Gadolinium injection reduced to 1/6th and the full dose sequences (Gold Standard). | 1 day

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU de Grenoble, Grenoble, Grenoble
  - CHU de Limoges, Limoges, Limoges
  - CHU de Lyon, Lyon, Lyon
  - CHU de Nantes, Nantes, Nantes
  - Fondation ophtalmique Adolphe de Rothschild, Paris, Paris
  - CHU de Rennes, Rennes, Rennes
  - CHU de Rouen, Rouen, Rouen
  - CHU de Strasbourg, Strasbourg, Strasbourg
  - CHU de Tours, Tours, Tours
  - CHU de Bordeaux, Bordeaux

IPD SHARING:
Plan to Share IPD: Undecided